CLINICAL TRIAL: NCT05602636
Title: Efficacy of Combined US-Guided Supraclavicular Block and Interscalene Analgesia Versus an Intercostobrachial Nerve Block Versus PCA With Fentanyl on Preventing Tourniquet Pain in Forearm Surgery: A Randomized Clinical Trial
Brief Title: Analgesic Effect of Supraclavicular Block and Interscalene Analgesia Versus an Intercostobrachial Nerve Block Versus PCA in Forearm Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of Clinical Pharmacy, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB 00012367-22-011-003
Record Dates: First submitted 2022-10-28; First posted 2022-11-02 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-07

CONDITIONS: Forearm Surgery; US-Guided Supraclavicular Block; Interscalene Analgesia; Tourniquet Pain
Keywords: Intercostobrachial Nerve Block; PCA with Fentanyl
MeSH Terms: interventions — Bupivacaine; Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- interscalene analgesia (Group ISBPB) (Active Comparator): All patients will receive a supraclavicular block as their primary anesthetic. Brachial plexus blocks will be performed at the supraclavicular fossa using 20 to 30 mL of 0.5% bupivacaine under ultrasound guidance.
  The C5 to C7 or C5 to C8 nerve roots between the anterior scalene and middle scalene muscles will be visualized in the absence of the subclavian artery and 10 mL 0.125% bupivacaine will be injected around the nerve roots of the brachial plexus. The needle trajectory will be adjusted to facilitate the even distribution of the local anesthetic around each nerve root.
  Interventions: Drug: bupivacaine, midazolam
- The intercostobrachial nerve block ( Group ICBN) (Active Comparator): All patients will receive a supraclavicular block as their primary anesthetic. Brachial plexus blocks will be performed at the supraclavicular fossa using 20 to 30 mL of 0.5% bupivacaine under ultrasound guidance.
  The ICBN block will be performed with 10 mL of 0.5% bupivacaine in the plane deep to the pectoralis minor and/or serratus anterior muscle over the second and third intercostal space.
  Interventions: Drug: bupivacaine, midazolam
- Patient-Controlled Analgesia (Group PCA) (Active Comparator): All patients will receive a supraclavicular block as their primary anesthetic. Brachial plexus blocks will be performed at the supraclavicular fossa using 20 to 30 mL of 0.5% bupivacaine under ultrasound guidance.
  Interventions: Drug: bupivacaine, midazolam

INTERVENTIONS:
Drug: bupivacaine, midazolam — Patients will be provided with midazolam (up to 2 mg) if requested. No opioids will be administered before the incision. At the first patient complaint of pain, the intraoperative anesthesia team will document the quality and location of pain, and 50 microgram of fentanyl will be administered if the patient requested it or pain score more than 3

SUMMARY:
The etiology of tourniquet pain is complex, and the study team hypothesizes that blocking with Interscalene brachial plexus block (ISBPB) is more efficient in decreasing the incidence of tourniquet pain in comparison with other techniques.

As there is a paucity of studies that evaluate the effect of intercostobrachial nerve (ICBN) block and ISBPB and Patient-Controlled Analgesia (PCA) with a supraclavicular brachial plexus block (SCBPB) on tourniquet pain in forearm surgery, Therefore, we established this randomized study to compare ISBPB and ICBN and PCA with fentanyl with SCBPB in terms of the incidence and severity of tourniquet pain in patients undergoing forearm surgery.

ELIGIBILITY:
Inclusion Criteria:

* aged more than 18 years,
* ASAI-III patients
* scheduled to undergo orthopedic or plastic surgery distal to the elbow with an anticipated tourniquet duration greater than 45 min.
* desiring regional anesthesia as the primary anesthetic.

Exclusion Criteria:

* Contraindication to regional anesthesia.
* Allergy to local anesthetics.
* Primary block failure.
* If patients desired deep intraoperative sedation.
* Clinically significant cognitive impairment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of tourniquet pain | 2 hours
  The incidence of tourniquet pain will be assessed by the patient's VAS score. The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). The patient is asked to rate their current level of pain by placing a mark on the line.

SECONDARY OUTCOMES:
Hemodynamics | 2 hours
  Hemodynamics up to 2 hours postoperative (heart rate, mean arterial blood pressure. Mean arterial blood pressure and heart rate will be recorded at baseline and every 5 min till the end of the procedure.
The incidence of adverse reactions | 2 hours
  The incidence of adverse reactions (Pneumothorax, Horner's syndrome) will be evaluated.
Patients' satisfaction | 24 hours
  Patients' satisfaction will be measured immediately postoperative and after 24 hours using a five-point Likert scale consisting of "very dissatisfied," "dissatisfied," "unsure," "satisfied," and "very satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Facualty of Medicine(Damietta), Al Azhar University, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared with a reasonable request from the corresponding auther
Supporting Information: Study Protocol, SAP